CLINICAL TRIAL: NCT06525662
Title: Randomised Controlled Trial of Stylet Shape in Simulated Endotracheal Intubation by Medical Students
Brief Title: Stylet Shape in Simulated Endotracheal Intubation by Medical Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NUS-L2023-08-01
Record Dates: First submitted 2024-07-08; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Endotracheal Intubation; Medical Education
Keywords: Medical education; Simulation

STUDY DESIGN:
Intervention Model Description: Design: Randomised controlled trial with 2 parallel groups Population: Final year medical students in NUS Medicine learning endotracheal intubation (ETI) with direct laryngoscopy using a Macintosh blade via simulation. These students have limited exposure to ETI and are novices in this procedure.
  Intervention: 30-degree STC styleted endotracheal tube (ETT) Comparator: Arcuate styleted ETT
Who Masked: Care Provider
Masking Description: The instructors teaching students how to use the different stylet shapes will be masked regarding the study hypothesis and participant group allocation. It will be emphasised to instructors that each participant has an equal amount of time to learn to use both shapes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30-degree straight to cuff (Experimental): The endotracheal tube to be used for endotracheal intubation will have a stylet inserted into it and manipulated into a shape that is straight from its proximal end to the cuff. At the cuff, there will be a 30 degree anterior bend.
  Interventions: Procedure: Endotracheal intubation using an endotracheal tube with a 30 degree straight to cuff shape
- Arcuate (Active Comparator): The endotracheal tube to be used for endotracheal intubation will have a stylet inserted into it and manipulated into an arcuate shape, and thus curved throughout the length of the tube.
  Interventions: Procedure: Endotracheal intubation using an endotracheal tube with an arcuate cuff shape

INTERVENTIONS:
Procedure: Endotracheal intubation using an endotracheal tube with a 30 degree straight to cuff shape — Placement of an endotracheal tube into a simulated trachea in a mannequin using the abovementioned shape
  Arms: 30-degree straight to cuff
Procedure: Endotracheal intubation using an endotracheal tube with an arcuate cuff shape — Placement of an endotracheal tube into a simulated trachea in a mannequin using the abovementioned shape
  Arms: Arcuate

SUMMARY:
Endotracheal intubation is a life saving procedure where a tube is placed into a person's windpipe to help them to breathe. This is a study of which shape of tube would lead to improved success in this procedure.

DETAILED DESCRIPTION:
Endotracheal intubation (ETI) is a lifesaving procedure. It involves placing a tube in the patient's airway to maintain ventilation and oxygenation.

Simulation has been shown to be effective for medical procedural skills training. Medical simulation literature now focuses on instructional design (ID) features that improve learning.

There are multiple aspects of ETI technique and ID that can be modified to improve successful ETI. Patient positioning, mastery learning, and dyad rather than solo practice are examples for which evidence exists to guide instructors. Despite this, ETI complication rates are substantial.

Thus, areas for continued improvement in ETI ID should be explored. One area is the optimal endotracheal tube (ETT) shape, achieved using a stylet, for novices learning ETI, for which there is limited evidence.

The straight to cuff (STC) shape has been postulated to optimise views of the airway compared to an arcuate shape. These shapes have only been directly compared as subgroups among multiple other comparisons in ETI technique in difficult intubations in one study. This does not generalise well to educating novices such as medical students, where intubations at normal difficulty are within the learner's zone of proximal development, and findings from subgroup comparisons are hypothesis generating rather than definitive evidence

This study will compare which shape is most likely to lead to successful endotracheal intubation, when performed by novices (medical students) learning this procedure on mannequins.

ELIGIBILITY:
Inclusion Criteria:

* Final year medical students in the Yong Loo Lin School of Medicine, National University of Singapore, undergoing their simulation posting. Endotracheal intubation is a procedure that is taught during this posting.

Exclusion Criteria:

* Injuries precluding performance of endotracheal intubation. Non exhaustive examples include arm injuries.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to successful intubation | Outcome assessment will occur within 2 weeks of endotracheal intubation being taught to participants, and immediately upon randomisation to a specified shape to attempt endotracheal intubation under video recording
  Defined as the time between insertion of the laryngoscope to successful placement of the tube in the trachea

SECONDARY OUTCOMES:
Proportion of participants who successfully intubate on first pass of laryngoscope | Outcome assessment will occur within 2 weeks of endotracheal intubation being taught to participants, and immediately upon randomisation to a specified shape to attempt endotracheal intubation under video recording
  Defined as successful placement of the tube into the trachea with only one insertion of the laryngoscope blade into the mouth
Proportion of participants who successfully intubate on first pass of endotracheal tube | Outcome assessment will occur within 2 weeks of endotracheal intubation being taught to participants, and immediately upon randomisation to a specified shape to attempt endotracheal intubation under video recording
  Defined as successful placement of the tube into the trachea with only one insertion of the endotracheal tube into the mouth
Proportion of participants who perform an oesophageal intubation | Outcome assessment will occur within 2 weeks of endotracheal intubation being taught to participants, and immediately after their intubation attempt under video recording
  Defined as placement of the endotracheal tube into the oesophagus as the end state of the participant's attempt

CONTACTS AND LOCATIONS:
Overall Officials: Matthew JW Low, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- Yong Loo Lin School of Medicine, National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
No plan for this, as this was not a part of the approved IRB application